CLINICAL TRIAL: NCT05579392
Title: Bright Light Therapy in Crohn's Disease on Intestinal Barrier Homeostasis
Brief Title: A Randomized Crossover Trial of Bright Light Therapy in Crohn's Disease on Intestinal Barrier Homeostasis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Ali Keshavarzian, Principle Investigator, Rush University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 22041302
Record Dates: First submitted 2022-09-22; First posted 2022-10-13 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Ultraviolet Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to receive Bright light therapy or placebo (wearing a similar device but will not receive the therapy) for 4 weeks, then they will do a washout period. After the washout period, the same participants will crossover to the opposite group for the remaining 4 weeks of the study, i.e. placebo or bright light therapy.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bright Light Therapy via ReTimer glasses, Then Placebo (Experimental): Participants will wear their device for 60 minutes every morning for 28-days (4 weeks)
  Interventions: Device: Bright Light Therapy; Device: Placebo Retimer Device
- No Bright Light Therapy via placebo glasses, Then Bright Light Therapy (Experimental): Participants will wear their placebo device for 60 minutes every morning for 28-days (4 weeks)
  Interventions: Device: Bright Light Therapy; Device: Placebo Retimer Device

INTERVENTIONS:
Device: Bright Light Therapy — Device: Bright Light Therapy Retimer
Device: Placebo Retimer Device — Device: Placebo Retimer Device with no bright light therapy

SUMMARY:
Crohn's Disease (CD) and Ulcerative Colitis (UC), collectively known as inflammatory bowel disease (IBD), are two of the most significant chronic conditions of the gastrointestinal tract (GIT) and affects over 1.5 million individuals in the U.S. Recently, there has been an increased understanding of the importance of sleep and sleep disruption in IBD as a potentially modifiable risk factor. We, therefore, hypothesize that intervening with morning bright light therapy (BLT) in IBD patients with CM will decrease intestinal permeability and pro-inflammatory cytokines, positively impact intestinal microbiota, and improve quality of life (QoL).

DETAILED DESCRIPTION:
Crohn's Disease (CD) and Ulcerative Colitis (UC), collectively known as inflammatory bowel disease (IBD), are two of the most significant chronic conditions of the gastrointestinal tract (GIT). IBD affects over 1.5 million individuals in the US, so identifying risk factors for disease flares is essential to avoid complications, such as hospitalizations and surgery, and to improve quality of life (QoL). Recently, there has been an increased understanding of the importance of sleep and sleep disruption in IBD as a potentially modifiable risk factor.

Bright light therapy (BLT) in IBD patients with CM may decrease intestinal permeability and pro-inflammatory cytokines, positively impact intestinal microbiota, and improve quality of life (QoL).In order to administer BLT efficiently and safely, a Re-Timer device, which is a lightweight, wearable set of glasses that emits blue-green light. Please note, the FDA has determined this device to be a General Wellness product and is not regulated by the FDA.

Prior to starting treatment, IBD patients will be screened for subclinical inflammation using a fecal calprotectin (FC) level and a blood test. If no subclinical inflammation is detected, potential subjects will be informed of their ineligibility. Eligible participants will complete questionnaires assessing their dietary habits, fatigue, sleep habits, quality of life, and severity of their underlying disease. Participants will also be provided a wrist actigraphy, which is a watch like device, to wear for 21 days to objectively assess CM prior to initiating therapy. Once the subjects demonstrate both subjective and objective evidence of CM, during their follow-up visit they will be randomly assigned to wear either the Re-Timer device to receive BLT or the placebo Re-Timer device (non BLT) for 4 weeks. Prior to and following receiving BLT or non BLT placebo, the following samples will be obtained: i) serum markers of inflammation and endotoxemia, ii) urine samples to test for intestinal permeability, and iii) stool samples to assess intestinal microbiota. These proposed studies will assess whether BLT has an impact on IBD patients' inflammation, intestinal permeability, and intestinal microbiota.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy proven diagnosis of Crohn's or Ulcerative Colitis
2. 18 years or older
3. Fecal Calprotectin > 50 or CRP above upper limit of normal or a PROMISE Fatigue ≥ 50
4. Has been on a stable dose of either a biologic, immunomodulator, or 5-ASA for at least 12 weeks

Exclusion Criteria:

1. Active IBD (Harvey Bradshaw Index > 5 or Modified Harvey Bradshaw Index >5)
2. Major depression (score ≥ 21 or any endorsement of suicidal intent on the Beck Depression)
3. Sleep apnea (score high risk in 2 or more categories of the Berlin Questionnaire) (43)
4. Restless leg syndrome (score ≥ 15 on the IRLS Study Group Rating Scale(44))
5. Regular use of medications that affect intestinal permeability, and/or endogenous melatonin including metoclopramide, NSAIDs, beta blockers, psychotropic medications, hypnotics and exogenous melatonin products during 4 weeks prior to the study
6. People who have worked night shifts or crossed more than 2 time zones in the previous month
7. Any major organ disease - renal impairment (creatinine>1.2 mg/dL), diabetes (Hgb-A1c > 6.5%); liver disease (LFTs > 1.5x normal), or significant cardiac failure (NY classification stage III/IV)
8. Diagnosis of narrow angle glaucoma or retinal disorders or demonstrated symptoms indicative of these diagnosis during the eligibility screening
9. Inability to sign an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-22 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Changes in intestinal permeability (% excretion of urinary sucralose) | 15 weeks
  Participants will ingest a sugar cocktail at Visits 2-5 and complete a urine collection. Measurement of urinary sugars is done using gas chromatography is used to calculate intestinal permeability.
Changes in microbiota will be assessed using shotgun metagene sequencing and total microbial community DNA | 15 weeks
  At all study visits, stool samples will be collected and analyzed using shotgun metagene sequencing and total microbial community DNA will be isolated and processed for microbiome analysis.

SECONDARY OUTCOMES:
Change in systemic markers of barrier disruption and inflammation | 15 weeks
  Inflammatory cytokines (IL-6, TNF-α, and IL-8) are the markers of disruption. IL-6, IL-8, and TNF-α will be measured in the plasma.
Change in systemic markers of inflammation | 15 weeks
  markers of endotoxemia (LPS, LBP, and sCD14) will be used to assess inflammation. Lipopolysaccharide binding protein(LBP) and sCD14 will be measured in serum by high sensitivity ELISA. Lipopolysaccharide (LPS) will be measured in serum using a LAL assay which is a quantitative, kinetic assay for the detection of Gram-negative bacterial endotoxin.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Keshavarzian, M.D., Principal Investigator — Rush University Medical Center; Garth R Swanson, M.D., Principal Investigator — Medical University of South Carolina
Locations (2):
- United States (2):
  - Rush University Medical Center, Chicago, Illinois
  - Medical University of South Carolina, Charleston, South Carolina